CLINICAL TRIAL: NCT05477797
Title: Id and Rd Maintenance Regimens After Induction of Remission in Multiple Myeloma: a Prospective, Randomized, Controlled, Multicenter Clinical Study
Brief Title: Id and Rd Maintenance Regimens After Induction of Remission in Multiple Myeloma.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-029-B
Record Dates: First submitted 2022-07-20; First posted 2022-07-28 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Progression Free Survival; Overall Survival; Maintenance
Keywords: multiple myeloma;; maintenance
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into two groups（Id，Rd）after risk stratification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ixazomib DX (Experimental): Id: Ixazomib 4mg po d1,8,15; Dexamethasone 20mg po d1,8,15,22; （28 days /cycle）. The treatment will be maintained for 2 years （if no disease progression or intolerant side effects appear）.
  Interventions: Drug: Ixazomib DX/Lenalidomide DX
- Lenalidomide DX (Placebo Comparator): Rd: Lenalidomide 25mg qd d1-21; Dexamethasone 20mg po d1,8,15,22; （28 days /cycle）. The treatment will be maintained for 2 years （if no disease progression or intolerant side effects appear）.
  Interventions: Drug: Ixazomib DX/Lenalidomide DX

INTERVENTIONS:
Drug: Ixazomib DX/Lenalidomide DX — After assessment of risk stratification，patients will be assigned to Id or Rd group randomly for maintenance therapy. Then they will be reviewed the efficacy monthly.
  Other Names: Id/Rd

SUMMARY:
Newly Diagnosed Myeloma Patients, who achieved efficacy above VGPR (very good PR)after initial treatment were enrolled. Patients were then randomly assigned to Id and Rd groups for maintenance treatment. Therapeutic effectiveness will be reviewed monthly until intolerant side effect or disease progression appear . The follow-up period is approximately 2 years.

DETAILED DESCRIPTION:
Newly Diagnosed Myeloma Patients, who achieved efficacy above VGPR after initial treatment were enrolled. Patients were then randomly assigned to Id and Rd groups for maintenance treatment. Therapeutic effectiveness will be reviewed monthly until intolerant side effect or disease progression appear . The follow-up period is approximately 2 years. Progression-free survival (PFS)was defined as the duration from randomization to the first evidence of disease progression or death from any cause. Overall survival (OS) was defined as the duration from the randomization to death from any cause. The Kaplan-Meier method was employed to plot the survival curves, with the log-rank test to assess the differences.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients aged 18 years or older with a confirmed diagnosis of symptomatic diagnosed multiple myeloma. Patients who have previously received initial treatment (induction, transplantation and consolidation are considered to be the same as first-line treatment) and the efficacy assessment ≥VGPR after the initial therapy.
2. An informed consent form (ICF) has been signed. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the disease, the legal guardian or the patient's immediate family will sign the informed consent;
3. Female patients of child-bearing potential should meet both of the following criteria:

   1. Take effective contraceptive measures during the study and for three months following the last dose;
   2. A negative serum pregnancy test at screening. Note: Women of childbearing potential include all the female who have started menstruating and are not post-menopausal and have not undergone surgical sterilization(eg, hysterectomy, double tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for more than 12 consecutive months due to unspecified reasons.
4. Male subjects(including those undergo vasectomy) agree to use condoms if sexually active with a female of child-bearing potential from the date of signing the informed consent. And no plan of pregnancy throughout the study and for three months following the last dose.
5. There are follow-up conditions. The patients known about the characteristics of the disease and voluntarily join the study program for treatment and follow-up.
6. Complete documentation of of the initial therapy is available.

   * Details of the state treatment and remission
   * cytogenetics at diagnosis
   * R-ISS staging at diagnosis
7. Eastern Cooperative Oncology Group Performance Status of 0 to 2.
8. Patient is willing and able to adhere to the study visit schedule and other protocol requirements including blood sampling and bone marrow aspiration.
9. Patients must meet the following clinical laboratory criteria at study entry:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3 without growth factor support. Platelet count ≥ 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before randomization.
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase and aspartate aminotransferase ≤ 3 x ULN.
   * Calculated creatinine clearance ≥ 30 mL/min (using the Cockcroft-Gault equation.

Exclusion Criteria:

1. Multiple myeloma that has relapsed after initial therapy.
2. Radiotherapy or major surgery within 14 days before randomization.
3. Diagnosed or treated for another malignancy within 1 years before randomization or previous diagnosis with another malignancy with evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
4. Infection requiring IV antibiotic therapy or other serious infection within 14 days before randomization.
5. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, uncontrolled congestive heart failure, unstable angina.
6. Systemic treatment with strong CYP3A inducers(rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) .
7. Ongoing or active infection, known human immunodeficiency virus positive, active hepatitis B or C infection.
8. Comorbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (e.g., PN of any cause that is Grade 1 with pain or Grade 2 or higher).
9. Psychiatric illness/social situation that would limit compliance with study requirements.
10. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
11. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or GI procedure that could interfere with the oral absorption or tolerance of treatment.
12. Treatment with any investigational products within 30 days before randomization.
13. Female patient who is lactating and breastfeeding or has a positive serum pregnancy test during the Screening period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
the percentage of 2 year PFS(progression-free survival) | from randomization to the end of 2years maintenance.
  the percentage of the patients whose disease do not appear progression at the end of 2years maintenance from each group.

SECONDARY OUTCOMES:
OS(overall survival) | from duration from the randomization to the end of 2years maintenance
  OS of the either group patients

OTHER OUTCOMES:
side effect | from randomization to the end of 2years maintenance
  side effect of each group within 2 years of maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Lu Zhong, Principal Investigator — RenJi Hospital
Locations (1):
- shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No